CLINICAL TRIAL: NCT01659827
Title: A Prospective, Randomized, Blinded, Comparative Study of Amniotic Membrane Injectable in the Treatment of Recalcitrant Plantar Fasciitis
Brief Title: Comparative Study of Amniotic Membrane Injectable in the Treatment of Recalcitrant Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIPF001
Record Dates: First submitted 2012-08-02; First posted 2012-08-08 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Control (Sham Comparator): Initial injections of Marcaine and Saline (one each)
  Interventions: Other: Marcaine; Other: Saline
- 0.5cc AmnioFix Injectable (Experimental): Initial injections of Marcaine and 0.5cc AmnioFix (one each)
  Interventions: Other: Marcaine; Other: 0.5cc AmnioFix
- 1.25cc AmnioFix Injectable (Experimental): Initial injections of Marcaine and 1.25cc AmnioFix (one each)
  Interventions: Other: Marcaine; Other: 1.25cc AmnioFix

INTERVENTIONS:
Other: Marcaine — Injection of 2cc of Marcaine
Other: 0.5cc AmnioFix — Injection of 0.5cc of AmnioFix Injectable
  Arms: 0.5cc AmnioFix Injectable
Other: 1.25cc AmnioFix — Injection of 1.25cc of AmnioFix Injectable
  Arms: 1.25cc AmnioFix Injectable
Other: Saline — Injection of 1.25cc of Saline
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether the AmnioFix Injectable human amniotic membrane is effective in the treatment of recalcitrant plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Both male and female patients will be selected.
3. Plantar fasciitis has been treated with conservative usual care for at least 8 weeks, including at least three of the following modalities

   1. RICE
   2. Corticosteroid injection
   3. Stretching exercises
   4. NSAIDs
   5. Orthotics
4. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
5. Patient understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
6. Patient has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

1. Prior surgery at the site
2. Site that exhibits clinical signs and symptoms of infection
3. History of chronic plantar fasciitis of more than twelve months
4. Evidence of significant neurological disease of the feet
5. Non Ambulatory Patients
6. The presence of comorbidities that can be confused with or can exacerbate the condition including:

   * Calcaneal stress fracture
   * Nerve entrapment syndrome (baxter nerve syndrome or tarsal tunnel)
   * Plantar fascial rupture
   * Systemic disorders associated with enthesiopathy such as Gout, Reiters syndrome, rheumatoid arthritis, etc.
   * Achilles tendonitis
   * Fat pad atrophy
   * Fibromyalgia
7. Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
8. Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding Screening.
9. History of radiation at the site.
10. Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
11. Study foot has been previously treated with tissue engineered materials such as PRP within the last 30 days.
12. Patients who are unable to understand the aims and objectives of the trial.
13. Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
14. Pregnant or breast feeding. No pregnancy within the past 6 months.
15. Allergy to Gentamycin Streptomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in American Orthopaedic Foot and Ankle Society (AOFAS) Hind Foot Score at 8 Weeks | 8 Weeks

SECONDARY OUTCOMES:
Time to return to normal activities | Up to 8 Weeks
Pain scale | Weekly up to 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Zelen, DPM, Principal Investigator — Professional Education and Research Institute
Locations (2):
- United States (2):
  - Professional Education and Research Institute, Roanoke, Virginia
  - Professional Education and Research Institute, Salem, Virginia